CLINICAL TRIAL: NCT06096311
Title: Improvement of Hyperglycemia/Diabetes in Patients to Improve Safety
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amisha Wallia, Associate Professor, Northwestern University
Other Study IDs: STU00090319
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Interviews — Interviews

SUMMARY:
The goal of this project is to bring together staff and clinicians from Northwestern University/Northwestern Medical Group/Northwestern Memorial Hospital as well as patients and caregivers to assess and redesign the identification and management of hyperglycemia and diabetes during and in transitions of care. There will be 3 different groups for the study: a group of providers [Group 1], a group of patients/caregivers and laypersons [Group 2], and a stakeholder group [Group 3]. Participants will be asked to provide input on potential interventions for a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Provider Group: Multidisciplinary clinical team (including but not limited to inpatient endocrine nurse practitioners, nurse coordinators, diabetes educators, outpatient nurses, attending physicians, and pharmacists)
* Patient, Caregiver and Layperson Group: Patients must have had hyperglycemia or diabetes at Northwestern Memorial Hospital in the last 5 years.
* Stakeholder Group: Involved in the specific care delivery of diabetes

Exclusion Criteria:

* Provider Group: None
* Patient, Caregiver, and Layperson Group: Patients will be excluded if they did not have diabetes or had hyperglycemia.
* Stakeholder Group: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Provider Group: A clinical multidisciplinary team including inpatient endocrine nurse practitioners, nurse coordinators, diabetes educators, outpatient nurses, attending physicians, and pharmacists.
  Patient, Caregiver and Layperson Group: The patients who have diabetes/hyperglycemia seen by the Glucose Management Service, the diabetes educator, or the endocrinology service. Caregivers will only be identified by patients if there was a member of their family who helped them with their diabetes management. Laypersons will be identified by research staff as members of the community that can directly advance research and solution development in the field.
  Stakeholder Group: Any and all stakeholders that are currently involved in the specific care delivery of diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative Results from Interviews | Up to one year
  Participants will be asked to provide their thoughts on potential interventions for a future clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No